CLINICAL TRIAL: NCT02509286
Title: Perioperative Chemotherapy (FLOT Protocol) Compared To Neoadjuvant Chemoradiation (CROSS Protocol) in Patients With Adenocarcinoma of the Esophagus
Brief Title: Perioperative Chemotherapy Compared To Neoadjuvant Chemoradiation in Patients With Adenocarcinoma of the Esophagus
Acronym: ESOPEC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Clinical Trials Unit Freiburg (Other); University of Freiburg (Other); University of Leipzig (Other); University of Luebeck (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Jens Hoeppner, Deputy Director - Department of Surgery, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P000760; 2015-001683-20 (EudraCT Number); DRKS00008008 (Registry Identifier: DRKS)
Record Dates: First submitted 2015-07-22; First posted 2015-07-28 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Adenocarcinoma (UICC TNM7); Adenocarcinoma of the Esophagogastric Junction
Keywords: Esophageal neoplasms; gastro-esophageal junction neoplasms; adenocarcinoma; esophagectomy; surgery; radiotherapy; chemotherapy
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Adenocarcinoma | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Carboplatin; Paclitaxel; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative Chemotherapy (FLOT): (Experimental): The FLOT Arm consists of the FLOT protocol, which consists of 5-Fluorouracil, Leucovorin, Oxaliplatin and Docetaxel. Repetition every 2 weeks (d15, q2w). Four neoadjuvant cycles (8 weeks) prior to surgery and four adjuvant cycles (8 weeks) postoperatively are given.
  Surgery is carried out by transthoracic subtotal esophagectomy or by transabdominal distal esophageal resection plus gastrectomy depending on tumor localization.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel
- Neoadjuvant Chemoradiation (CROSS): (Active Comparator): The CROSS Arm consists of the CROSS protocol, which consists of neoadjuvant radiation therapy (41.4Gy / 23fractions) and concurrent chemotherapy with Carboplatin and Paclitaxel (5 weeks) prior to surgery.
  Surgery is carried out by transthoracic subtotal esophagectomy or by transabdominal distal esophageal resection plus gastrectomy depending on tumor localization.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Neoadjuvant radiation

INTERVENTIONS:
Drug: 5-Fluorouracil — 2600 mg/m² (24 hours), d1 every two weeks;
  Arms: Perioperative Chemotherapy (FLOT):
Drug: Leucovorin — 200 mg/m² in 250 ml NaCl 0.9%, d1 every two weeks;
  Arms: Perioperative Chemotherapy (FLOT):
Drug: Oxaliplatin — 85 mg/m² in 500 ml G5% over 2h, d1 every two weeks;
  Arms: Perioperative Chemotherapy (FLOT):
Drug: Docetaxel — 50mg/m2 in 250 ml NaCl 0.9% over 1h, d1 every two weeks;
  Arms: Perioperative Chemotherapy (FLOT):
Drug: Carboplatin — Dose-dependant: 2mg/ml/min AUC in 500ml Glucose 5%, day 1, 8, 15, 22 and day 29.
  Arms: Neoadjuvant Chemoradiation (CROSS):
Drug: Paclitaxel — 50mg/m2 in 500ml NaCl 0.9% over 1 h, day 1, 8, 15, 22 and day 29;
  Arms: Neoadjuvant Chemoradiation (CROSS):
Radiation: Neoadjuvant radiation — 41.4Gy given in 23 fractions of 1.8Gy on days 1-5, days 8-12, days 15-19, days 22-26 and days 29-31.
  Arms: Neoadjuvant Chemoradiation (CROSS):

SUMMARY:
The trial is designed to investigate differences in outcome of patients with esophageal adenocarcinoma and junctional adenocarcinoma treated with perioperative (neoadjuvant + adjuvant) chemotherapy (FLOT) plus surgical resection versus neoadjuvant chemoradiation (CROSS) plus surgical resection.

DETAILED DESCRIPTION:
According to the given evidence a survival benefit of perioperative chemotherapy (periCTX) over Neoadjuvant chemoradiation (neoCRT) for patients with Esophageal adenocarcinomas (EAC) has not been proven in any randomized controlled trials (RCT). Data supporting the value of periCTX have all been obtained in studies including mixed patient cohorts with EAC and gastric adenocarcinoma (GAC). Due to relevant differences of histologic subtype distribution, response to periCTX and survival rates between EAC and GAC there is a clear need to obtain evidence concerning the value of periCTX for EAC. As nowadays periCTX is extensively and successfully applied in clinical practice in patients with EAC there is an obvious need to obtain evidence from a multicentre RCT. Moreover a confirmation of the superior survival rates of the recent RCT on neoCRT should be obtained in a RCT conducted exclusively on EAC. Therefore, this prospective RCT with the primary objective of longterm patient survival comparing periCTX and neoCRT was designed.

Translational Projects:

Project 1+2: Circulating Tumor Cells as Biomarker in EAC CTC laboratories at University of Hamburg and University of Freiburg Project 3: Prognostic and predictive biomarkers in EAC University of Leipzig, UCCL

ELIGIBILITY:
Inclusion criteria:

* Histologically verified adenocarcinoma of the esophagus according to the UICC definition (TNM7)
* Pre-treatment stage cT1N+, M0 or cT2-4a, N0/+, M0
* Age ≥18 years
* No prior abdominal or thoracic radiotherapy
* ECOG Performance status 0-2
* Adequate cardiac function ( Patients with a cardiac history (e.g. myocardial infarction, heart failure, coronary artery disease) should have a cardiology review)
* Adequate bone marrow function (WBC>3x10^9/l; Hb>9g/dl; platelets >100x10^9/l)
* Adequate respiratory function. Symptomatic Patients should have pulmonary function tests with FEV1 >65% of predicted)
* Adequate renal function (GFR >60ml/min)
* Adequate liver function (serum bilirubin <1.5x Upper level of Normal (ULN); AST <2.5x ULN and ALT <3x ULN (ULN as per institutional standard)
* written informed consent

Exclusion Criteria:

* Tumors of squamous or other non-adenocarcinoma histology
* Patients with advanced inoperable or metastatic esophageal adenocarcinoma
* Stage cT1N0 and cT4b
* Gastric carcinoma
* Prior chemotherapy for cancer,
* Clinically significant (i.e. active) cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months)
* Clinical significant lung disease (FEV1 <65% of predicted)
* Peripheral neuropathy Grade >1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2016-01; Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At end of trial- up to 3 years in follow up
  Overall survival will be calculated as time from start of study treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival time (PFS) | From randomisation up to 3 years in follow up
  PFS will be calculated as the time interval from randomisation to the first event of locoregional failure, metastatic progression or death.
Site of failure: local, regional or distant Failure | From time of surgery up to 3 years in follow up
Recurrence free survival time | From time of surgery up to 3 years in follow up
  RFS will be calculated in resected patients who achieved an R0 or R1 resection as the time interval from surgery to the date of first recurrence (local, regional or distant) or death, whatever comes first.
Postsurgical Quality of Life | From randomization up to 3 years in follow up
Postoperative complications | From time of surgery up to 90 days postoperatively
Non-surgical site complications | From time of surgery up to 90 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hoeppner, Professor, Principal Investigator — University Medical Center Schleswig-Holstein, Campus Lübeck
Locations (30):
- Germany (30):
  - Uniklinik RWTH Aachen, Aachen
  - Charité Berlin - Campus Benjamin Franklin (CBF), Berlin
  - Charité Berlin Campus Virchow-Klinikum (CVK), Berlin
  - Uniklinik Köln, Cologne
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München (LMU), München
  - Universitätsklinikum Münster, Münster
  - Ruppiner Kliniken GmbH, Neuruppin
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsmedizin Rostock, Rostock
  - Klinikum Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - Klinikum Mutterhaus, Trier
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Background] Hoeppner J, Lordick F, Brunner T, Glatz T, Bronsert P, Rothling N, Schmoor C, Lorenz D, Ell C, Hopt UT, Siewert JR. ESOPEC: prospective randomized controlled multicenter phase III trial comparing perioperative chemotherapy (FLOT protocol) to neoadjuvant chemoradiation (CROSS protocol) in patients with adenocarcinoma of the esophagus (NCT02509286). BMC Cancer. 2016 Jul 19;16:503. doi: 10.1186/s12885-016-2564-y. PMID 27435280
- [Derived] Hoeppner J, Brunner T, Schmoor C, Bronsert P, Kulemann B, Claus R, Utzolino S, Izbicki JR, Gockel I, Gerdes B, Ghadimi M, Reichert B, Lock JF, Bruns C, Reitsamer E, Schmeding M, Benedix F, Keck T, Folprecht G, Thuss-Patience P, Neumann UP, Pascher A, Imhof D, Daum S, Strieder T, Krautz C, Zimmermann S, Werner J, Mahlberg R, Illerhaus G, Grimminger P, Lordick F. Perioperative Chemotherapy or Preoperative Chemoradiotherapy in Esophageal Cancer. N Engl J Med. 2025 Jan 23;392(4):323-335. doi: 10.1056/NEJMoa2409408. PMID 39842010
- See also: ESOPEC Homepage — https://www.uniklinik-freiburg.de/esopec-studie.html